CLINICAL TRIAL: NCT03274492
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial Comparing the Efficacy and Safety of Polatuzumab Vedotin in Combination With Rituximab and CHP (R-CHP) Versus Rituximab and CHOP (R-CHOP) in Previously Untreated Patients With Diffuse Large B-Cell Lymphoma
Brief Title: A Study Comparing the Efficacy and Safety of Polatuzumab Vedotin With Rituximab-Cyclophosphamide, Doxorubicin, and Prednisone (R-CHP) Versus Rituximab-Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in Participants With Diffuse Large B-Cell Lymphoma
Acronym: POLARIX
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GO39942; 2017-002023-21 (EudraCT Number)
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- R-CHP plus Vincristine Placebo plus Polatuzumab Vedotin (Experimental): Participants will receive polatuzumab vedotin 1.8 milligrams per kilogram (mg/kg) intravenously (IV), placebo for vincristine IV, rituximab 375 milligrams per square meter (mg/m^2) IV, cyclophosphamide 750 mg/m^2 IV, and doxorubicin 50 mg/m^2 IV on Day 1 and prednisone 100 milligrams per day (mg/day) orally (PO) on Days 1-5 of every 21-day cycle for 6 cycles. Rituximab 375 mg/m^2 IV will be administered as monotherapy in Cycles 7 and 8.
  Interventions: Drug: Polatuzumab Vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine Placebo; Drug: Prednisone
- R-CHOP plus Polatuzumab Vedotin Placebo (Placebo Comparator): Participants will receive placebo for polatuzumab vedotin, rituximab 375 mg/m^2 IV, cyclophosphamide 750 mg/m^2 IV, doxorubicin 50 mg/m^2 IV, and vincristine 1.4 mg/m^2 IV (maximum 2 milligrams per dose [mg/dose]) on Day 1 and prednisone 100 mg/day PO on Days 1-5 of every 21-day cycle for 6 cycles. Rituximab 375 mg/m^2 IV will be administered as monotherapy in Cycles 7 and 8.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Polatuzumab vedotin Placebo

INTERVENTIONS:
Drug: Polatuzumab Vedotin — Polatuzumab vedotin IV infusion will be administered as per the schedule specified in the respective arm.
  Other Names: DCDS4501A; anti-CD79b-VC-MMAE
  Arms: R-CHP plus Vincristine Placebo plus Polatuzumab Vedotin
Drug: Rituximab — Rituximab IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Cyclophosphamide — Cyclophosphamide IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Doxorubicin — Doxorubicin IV infusion will be administered as per the schedule specified in the respective arm.
Drug: Vincristine — Vincristine IV infusion will be administered as per the schedule specified in the respective arm.
  Arms: R-CHOP plus Polatuzumab Vedotin Placebo
Drug: Vincristine Placebo — Placebo matching to vincristine will be administered as per the schedule specified in the respective arm.
  Arms: R-CHP plus Vincristine Placebo plus Polatuzumab Vedotin
Drug: Prednisone — Prednisone PO will be administered as per the schedule specified in the respective arm.
Drug: Polatuzumab vedotin Placebo — Placebo matching to polatuzumab vedotin will be administered as per the schedule specified in the respective arm.
  Arms: R-CHOP plus Polatuzumab Vedotin Placebo

SUMMARY:
This Phase III, randomized, double-blind, placebo-controlled study will compare the efficacy, safety, and pharmacokinetics of polatuzumab vedotin plus R-CHP versus R-CHOP in participants with previously untreated diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated participants with cluster of differentiation 20 (CD20)-positive DLBCL, including one of the following diagnoses by 2016 World Health Organization (WHO) classification of lymphoid neoplasms: DLBCL, not otherwise specified (NOS) including germinal center B-cell type, activated B-cell type; T-cell/histiocyte-rich large B-cell lymphoma; Epstein-Barr virus-positive DLBCL, NOS; anaplastic lymphoma kinase (ALK)-positive large B-cell lymphoma; human herpesvirus-8 (HHV8)-positive DLBCL, NOS; High-grade B-cell lymphoma with MYC and B-cell lymphoma 2 (BCL2) and/or B-cell lymphoma 6 (BCL6) rearrangements (double-hit or triple-hit lymphoma); High-grade B-cell lymphoma, NOS
* Availability of archival or freshly collected tumor tissue before study enrolment
* International Prognostic Index (IPI) score of 2-5
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Life expectancy greater than or equal to (>/=)12 months
* Left ventricular ejection fraction (LVEF) >/= 50 percent (%) on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
* Adequate hematologic function
* Female participants: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods and refrain from donating eggs.
* Male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom and agreement to refrain from donating sperm.

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Contraindication to any of the individual components of CHOP, including prior receipt of anthracyclines
* Prior organ transplantation
* Current Grade greater than (>) 1 peripheral neuropathy by clinical examination
* Demyelinating form of Charcot-Marie-Tooth disease
* History of indolent lymphoma
* History of follicular lymphoma grade 3B
* B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma (grey-zone lymphoma)
* Primary mediastinal (thymic) large B-cell lymphoma
* Burkitt lymphoma
* Prior treatment with cytotoxic drugs within 5 years of screening for any condition (example [e.g.], cancer, rheumatoid arthritis) or prior use of any anti-CD20 antibody
* Prior use of any monoclonal antibody within 3 months of the start of Cycle 1
* Prior therapy for DLBCL, with the exception of nodal biopsy
* Corticosteroid use >30 mg/day of prednisone or equivalent, for purposes other than lymphoma symptom control
* Participants with central nervous system (CNS) lymphoma (primary or secondary involvement), primary effusion DLBCL, and primary cutaneous DLBCL
* Vaccination with live vaccines within 28 days prior to the start of Cycle 1
* Any investigational therapy within 28 days prior to the start of Cycle 1
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Evidence of significant, uncontrolled, concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease or pulmonary disease
* Recent major surgery (within 4 weeks prior to the start of Cycle 1), other than for diagnosis
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third-degree heart block, or evidence of prior myocardial infarction
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or significant infections within 2 weeks before the start of Cycle 1
* Clinically significant liver disease, including active viral or other hepatitis, current alcohol abuse, or cirrhosis
* Prior radiotherapy to the mediastinal/pericardial region
* Participants with suspected active or latent tuberculosis
* Positive test results for chronic hepatitis B and hepatitis C infection
* Known history of human immunodeficiency virus (HIV) seropositive status
* Positive results for the human T-lymphotrophic 1 virus (HTLV-1)
* Participants with a history of progressive multifocal leukoencephalopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as Assessed by the Investigator, Using the Lugano Response Criteria for Malignant Lymphoma | From randomization to the first occurrence of disease progression or relapse, or death from any cause, whichever occurs earlier (up to 38 months)

SECONDARY OUTCOMES:
Percentage of Participants With Complete Response (CR) as Assessed by Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) by Blinded Independent Central Review (BICR) | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 8 [Cycle length=21 days] [up to Week 32])
Event-Free Survival-Efficacy (EFSeff) as Assessed by the Investigator, Using the Lugano Response Criteria for Malignant Lymphoma | From randomization to first occurrence of disease progression/relapse;or death from any cause;or other primary efficacy reason that leads to initiation of any non-protocol specified antilymphoma treatment(NALT);or residual disease(up to approx 65 months)
Percentage of Participants Who are Progression Free as Assessed by the Investigator, Using the Lugano Response Criteria for Malignant Lymphoma | 24 months after enrollment (up to approximately 65 months)
Overall Survival | From randomization until death from any cause (up to approximately 65 months)
Percentage of Participants With CR as Assessed by FDG-PET by Investigator | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 8 [Cycle length=21 days] [up to Week 32])
Disease-Free Survival (DFS) as Assessed by the Investigator, Using the Lugano Response Criteria for Malignant Lymphoma | From the date of first occurrence of a documented CR to the date of relapse or death from any cause (up to approximately 65 months)
Duration of Response as Assessed by the Investigator, Using the Lugano Response Criteria for Malignant Lymphoma | From the date of first occurrence of a documented CR or partial response (PR) to the date of progression, relapse, or death from any cause (up to approximately 65 months)
Event-Free Survival-All Causes (EFSall) as Assessed by the Investigator, Using the Lugano Response Criteria for Malignant Lymphoma | From randomization to disease progression or relapse, or death from any cause, or initiation of any NALT (up to approximately 65 months)
Time to Deterioration in European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30) Physical Functioning and Fatigue | Day 1 of Cycles 1, 2, 3 and 5 (Cycle length=21 days); treatment completion visit (TCV)/early treatment termination visit (ETTV) (up to approximately 32 weeks); post-treatment follow-up (FU) visit (up to approximately 65 months)
Time to Deterioration in Functional Assessment of Cancer Therapy-Lymphoma Lymphoma Subscale (FACT-Lym LymS) | Day 1 of Cycles 1, 2, 3 and 5 (Cycle length=21 days); TCV/ETTV (up to approximately 32 weeks); post-treatment FU visit (up to approximately 65 months)
Percentage of Participants Achieving Meaningful Improvement in EORTC QLQ-C30 Physical Functioning and Fatigue | Day 1 of Cycles 1, 2, 3 and 5 (Cycle length=21 days); TCV/ETTV (up to approximately 32 weeks); post-treatment FU visit (up to approximately 65 months)
Percentage of Participants Achieving Meaningful Improvement in FACT-Lym LymS | Day 1 of Cycles 1, 2, 3 and 5 (Cycle length=21 days); TCV/ETTV (up to approximately 32 weeks); post-treatment FU visit (up to approximately 65 months)
EORTC QLQ-C30 Treatment-Related Symptoms Score | Day 1 of Cycles 1, 2, 3 and 5 (Cycle length=21 days); TCV/ETTV (up to approximately 32 weeks); post-treatment FU visit (up to approximately 65 months)
Functional Assessment of Cancer Treatment/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-NTX) Peripheral Neuropathy Score | Day 1 of Cycles 1-8 (Cycle length=21 days); TCV/ETTV (up to approximately 32 weeks); post-treatment FU visit (up to approximately 65 months)
Percentage of Participants With adverse Events (AEs) | From randomization to the end of study (up to approximately 65 months)
Serum Concentration of Total Polatuzumab Vedotin | Pre-infusion (0 hour [hr]), 0.5 hr post-infusion (infusion duration=90 minutes [min]) on Day 1 of Cycle 1 and 4 (Cycle length=21 days); TCV/ETTV (up to approximately 32 weeks); post-treatment FU visit (up to approximately 65 months)
Plasma Concentration of Polatuzumab Vedotin Conjugate (Antibody-Conjugated Mono-Methyl Auristatin E [acMMAE]) | 0.5 hr post-infusion (infusion duration=90 min) on Day 1 of Cycle 1 and 4 (Cycle length=21 days); TCV/ETTV (up to approximately 32 weeks); post-treatment FU visit (up to approximately 65 months)
Plasma Concentration of Polatuzumab Vedotin Unconjugated MMAE | 0.5 hr post-infusion (infusion duration=90 min) on Day 1 of Cycle 1 and 4 (Cycle length=21 days); TCV/ETTV (up to approximately 32 weeks); post-treatment FU visit (up to approximately 65 months)
Percentage of Participants With Anti-Drug Antibody (ADA) to Polatuzumab Vedotin | Pre-infusion (0 hr) on Day 1 of Cycle 1 and 4 (Cycle length=21 days); TCV/ETTV (up to approximately 32 weeks); post-treatment FU visit (up to approximately 65 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (215):
- United States (50):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Southern Cancer Center, Daphne, Alabama
  - City of Hope, Duarte, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Rocky Mountain Cancer Centers, LLP, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Fort Myers (New Hampshire Ct), Fort Myers, Florida
  - Florida Cancer Specialists & Research Institute, St. Petersburg, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - University of Louisville Hospital, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center - Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center at Westchester, Harrison, New York
  - New York University Cancer Cen, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Levine Cancer Institute - Clincal Trials Administration, Charlotte, North Carolina
  - Oncology/Hematology Care Clinical Trials LLC, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oncology Associates of Oregon, P.C, Eugene, Oregon
  - Northwest Cancer Specialists - Portland (SW Barnes Rd), Portland, Oregon
  - Oregon HSU, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina Hospital, Charleston, South Carolina
  - Prisma Health ? Upstate, Greenville, South Carolina
  - Greco-Hainesworth Centers for Research, Chattanooga, Tennessee
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Oncology Associates of Southwest Virginia, Inc., Blacksburg, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia Uni Med. Center - Robert Byrd Health Science, Morgantown, West Virginia
- Australia (10):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital Woolloongabba, Woolloongabba, Queensland
  - Ashford Cancer Center Research, Kurralta Park, South Australia
  - The University of Adelaide - The Queen Elizabeth Hospital (TQEH), Woodville South, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
- Austria (3):
  - Paracelsus Medizinischen Privatuniversitaet-Salzburger Landeskliniken (SALK), Salzburg
  - Medizinische Universität Wien, Vienna
  - Wiener Gesundheitsverbund ? Klinik Ottakring, Vienna
- Belgium (3):
  - UZ Gent, Ghent
  - CH Jolimont - Lobbes (Jolimont), Haine-Saint-Paul
  - CHU UCL Mont-Godinne, Mont-godinne
- Brazil (4):
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Centro de Hematologia e Hemoterapia - HEMOCENTRO UNICAMP, Campinas, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Canada (7):
  - University of Alberta Hospital, Edmonton, Alberta
  - BC Cancer ? Vancouver, Vancouver, British Columbia
  - CancerCare Manitoba (CCMB), Winnipeg, Manitoba
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CIUSSS de l Est de l Ile de Montreal - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec
- China (13):
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - Jiangsu Cancer Hospital, Nanjing
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai East Hospital, Tongji University, Shanghai
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin
  - Tianjin Medical University Cancer Institute & Hospital, Tianjing
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou
- Czechia (5):
  - Fakultni Nemocnice Hradec Kralove (FNHK), Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Fakultni Nemocnice Kralovske Vinohrady (FNKV), Prague
  - Všeobecná fakultní nemocnice v Praze, Prague
- France (38):
  - CHU Amiens - Hopital Sud, Amiens
  - CHU Angers, Angers
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Institut d'Hématologie de Basse Normandie, Caen
  - CH Metropole de Savoie, Chambéry
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon - Hopital le Bocage, Dijon
  - L'Union Mutualiste de la Gestion des Eaux Claires - Institut Daniel Hollard, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Hôpital Albert Michallon, La Tronche
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
  - Hôpital Saint Vincent de Paul, Lille
  - Hopital Claude Huriez, Lille
  - Hopital Uni Ire Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - CHU Montpellier - Saint ELOI, Montpellier
  - CHU de Nantes - Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU de Nîmes - Hôpital Carémeau, Nîmes
  - Hôpital Saint-Louis, Paris
  - Gh Necker Enfants Malades, Paris
  - Hopital Saint Jean, Perpignan
  - Hopital Haut-Leveque - Centre Francois Magendie, Pessac
  - CHU Lyon Sud - Service Hématologie, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Centre Hospitalier de Quimper Cornouaille (CHIC), Quimper
  - Hopital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier de Saint Brieuc - Hôpital Yves Le Foll, Saint-Brieuc
  - Pôle de Cancérologie ? CHU de Saint?Etienne', Saint-Priest-en-Jarez
  - Chru de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer - Oncopole Toulouse (IUCT-O), Toulouse
  - CHU Bretonneau, Tours
  - CHU de Brabois, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique, Vannes
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Vivantes Klinikum Am Urban, Berlin
  - Städtisches Klinikum Dessau, Dessau
  - Universitätsklinikum Essen, Essen
  - Universitaetsklinikum Halle (Saale), Halle
  - Universitaetsklinikum Heidelberg, Heidelberg
  - InVO - Institut für Versorgungsforschung in der Onkologie GbR, Koblenz
  - Universitatsklinikum Munster, Münster
- Italy (8):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, Abruzzo
  - Universita degli Studi Di Brescia - Azienda Ospedaliera Spedali Civili di Brescia, Brescia, Abruzzo
  - Universita degli Studi di Roma ''La Sapienza" - Clinica Ematologica, Rome, Abruzzo
  - AUSL di Reggio Emilia, IRCCS, P.O. Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - IRCCS AOU San Martino - IST, Genoa, Liguria
  - Istituto Nazionale dei Tumori, Monza, Lombardy
  - Azienda Ospedaliero Universitaria Maggiore della Carita di Novara, Novara, Piedmont
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Turin, Piedmont
- Japan (19):
  - Aichi Cancer Center, Aichi
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital East, Chiba
  - Chiba University Hospital, Chūōku
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Hokkaido University Hospital, Hokkaido
  - Kobe City Medical Center General Hospital, Hyōgo
  - Tokai University Hospital, Isehara-shi
  - Kumamoto University Hospital, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Tohoku University Hospital, Miyagi
  - Osaka Metropolitan University Hospital, Osaka
  - The University of Osaka Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Jichi Medical University Hospital, Tochigi
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- New Zealand (3):
  - Auckland City Hospital, Cancer and Blood Research, Auckland
  - Canterbury Health Laboratories, Christchurch
  - Waikato Hospital, Hamilton
- Poland (5):
  - Samodzielny Publiczny Zak?ad Opieki Zdrowotnej Zespó? Szpitali Miejskich w Chorzowie, Chorzów
  - PRATIA MCM Kraków, Krakow
  - Uniwersytet Medyczny w Lodzi, Lodz
  - SPZOZ Ministerstwa Spraw Wewn?trznych i Administracji w Poznaniu, Późna
  - Wojskowy Instytut Medyczny - Panstwowy Instytut Badawczy, Warsaw
- Leningrad Regional Clinical Hospital, Saint Petersburg, Sankt-Peterburg, Russia
- South Korea (7):
  - Pusan National University Hospital, Busan
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (12):
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Catala d Oncologia Hospitalet, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitari Dr. Josep Trueta, Girona
  - Hospital Universitario La Paz, Madrid
  - Fundación Jimenez Díaz, Madrid
  - Hospital Quiron Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
- Universitätsspital Basel Gynäkologie - Onkologie, Basel, Switzerland
- Taiwan (5):
  - Kaohsiung Medical University Hospital, Cancer Center, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi-Mei Hospital, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (3):
  - Ankara University Faculty of Medicine Cebeci Hospital, Ankara
  - Ege Üniversitesi Tip Fakültesi, Lzmir
  - Dokuz Eylul Universitesi Tip Fakultesi, Lzmir
- Ukraine (3):
  - Communal Institution 'Cherkassy Regional Oncology Dispensary' of the Cherkassy Regional Council, Cherkassy, Chernihiv Governorate
  - MNE Lviv Territorial Medical Association Clinical Hospital for Palliative Care, Lviv, Chernihiv Governorate
  - Khmelnytskyi Regional Hospital, Khmelnytskyi, Kharkiv Governorate
- United Kingdom (8):
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrookes Hospital, Cambridge
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - University Hospitals of Leicester NHS Trust - Leicester Royal Infirmary, Leicester
  - Barts Health NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust. Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Thompson C, Trneny M, Morschhauser F, Salles G, Reagan PM, Hertzberg M, Zhang H, Thieblemont C, Hu B, Fonseca G, Kim WS, Martelli M, Mehta A, Singh A, Yan M, Hirata J, Sugidono M, Lee C, Sharman JP, Mehta-Shah N, Flowers CR, Tilly H, Chua N, Casasnovas RO, Miall F, Kim TM, Tsai XC, Nasta S, Lee ST, Friedberg JW. PROs vs clinician-reported adverse events in a large clinical trial: findings from the phase 3 POLARIX study. Blood. 2026 Jan 15;147(3):254-265. doi: 10.1182/blood.2025028848. PMID 40997297
- [Derived] Morschhauser F, Salles G, Sehn LH, Herrera AF, Friedberg JW, Trneny M, Lenz G, Sharman JP, Herbaux C, Burke JM, Matasar M, Collins GP, Mehta-Shah N, Oberic L, Chauchet A, Jurczak W, Song Y, Pinto A, Rai S, Izutsu K, Greil R, Mykhalska L, Bergua-Burgues JM, Cheung MC, Shin HJ, Hapgood G, Munhoz E, Abrisqueta P, Gau JP, Jiang Y, McCall B, Chohan S, Sugidono M, Yan M, Batlevi CL, Tilly H, Flowers CR. Five-Year Outcomes of the POLARIX Study Comparing Pola-R-CHP and R-CHOP in Patients With Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2025 Dec 10;43(35):3698-3705. doi: 10.1200/JCO-25-00925. Epub 2025 Sep 24. PMID 40991874
- [Derived] Hu B, Reagan PM, Sehn LH, Sharman JP, Hertzberg M, Zhang H, Kim A, Herbaux C, Molina L, Maruyama D, Stenner F, Chohan S, Kothari R, Lee Batlevi C, Hirata J, Sahin D, Lee C, Sugidono M, Tilly H. Subgroup analysis of older patients >/=60 years with diffuse large B-cell lymphoma in the phase 3 POLARIX study. Blood Adv. 2025 May 27;9(10):2489-2499. doi: 10.1182/bloodadvances.2024014707. PMID 40085955
- [Derived] Liao MZ, Deng R, Gibiansky L, Lu T, Agarwal P, Dere R, Lee C, Hirata J, Herbaux C, Salles G, Li C, Miles D. Ethnic sensitivity assessment: Polatuzumab vedotin pharmacokinetics in Asian and non-Asian patients with previously untreated diffuse large B-cell lymphoma in POLARIX. Clin Transl Sci. 2023 Dec;16(12):2744-2755. doi: 10.1111/cts.13669. Epub 2023 Oct 31. PMID 37864313
- [Derived] Song Y, Tilly H, Rai S, Zhang H, Jin J, Goto H, Terui Y, Shin HJ, Kim WS, Cao J, Feng J, Eom HS, Kim TM, Tsai XC, Gau JP, Koh H, Zhang L, Song Y, Yang Y, Li W, Huang H, Ando K, Sharman JP, Sehn LH, Bu L, Wang X, Jiang Y, Hirata J, Lee C, Zhu J, Izutsu K. Polatuzumab vedotin in previously untreated DLBCL: an Asia subpopulation analysis from the phase 3 POLARIX trial. Blood. 2023 Apr 20;141(16):1971-1981. doi: 10.1182/blood.2022017734. PMID 36626583
- [Derived] Varma G, Wang J, Diefenbach C. Polatuzumab vedotin in relapsed / refractory aggressive B-cell lymphoma. Expert Rev Anticancer Ther. 2022 Aug;22(8):795-803. doi: 10.1080/14737140.2022.2093191. Epub 2022 Jun 27. PMID 35726803
- [Derived] Tilly H, Morschhauser F, Sehn LH, Friedberg JW, Trneny M, Sharman JP, Herbaux C, Burke JM, Matasar M, Rai S, Izutsu K, Mehta-Shah N, Oberic L, Chauchet A, Jurczak W, Song Y, Greil R, Mykhalska L, Bergua-Burgues JM, Cheung MC, Pinto A, Shin HJ, Hapgood G, Munhoz E, Abrisqueta P, Gau JP, Hirata J, Jiang Y, Yan M, Lee C, Flowers CR, Salles G. Polatuzumab Vedotin in Previously Untreated Diffuse Large B-Cell Lymphoma. N Engl J Med. 2022 Jan 27;386(4):351-363. doi: 10.1056/NEJMoa2115304. Epub 2021 Dec 14. PMID 34904799